CLINICAL TRIAL: NCT05965349
Title: Evaluation of a Mindfulness-based Intervention on Depression Among Older Korean American Adults
Brief Title: MBCT Intervention: Healthy Mind, Healthy Living
Acronym: HMHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Asian American Resource and Information Network, Inc. (Other)
Responsible Party: Principal Investigator, Linda Ko, Professor: School of Public Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00015538
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Mindfulness Based Cognitive Therapy; Depression; Sleep; Anxiety Depression
Keywords: Mindfulness Based Cognitive Therapy (MBCT); Korean Americans; Group-based; Depression; Sleep
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group-based MBCT (Experimental): A telephone-based, 8-week MBCT session including: (1) learning mindfulness skills; (2) practicing mindfulness skills in class and at home; and (3) dialogue and inquiry.
  Interventions: Behavioral: Healthy Mind, Healthy Living

INTERVENTIONS:
Behavioral: Healthy Mind, Healthy Living — A telephone, 8-week MBCT workshop series including: (1) learning mindfulness skills; (2) practicing mindfulness skills in class and at home; and (3) dialogue and inquiry.

SUMMARY:
Depression among older Korean Americans are rising. Mindfulness-based cognitive therapy (MBCT) is an evidence-based intervention (EBI), effective for preventing depression relapse and reducing depressive symptoms. To enhance feasibility, acceptability, and reach, a brief version of MBCT has been developed and delivered by telephone (brief MBCT-T), but has only been tested in primarily White samples. This study will test test the effect of brief MBCT-T among older Korean Americans.

DETAILED DESCRIPTION:
Older Asians with limited English proficiency have experienced the greatest increase in depression before and during the COVID-19 pandemic compared to Whites, Blacks, and Hispanics. Social distancing measures to lower the risk of exposure to COVID-19, a diminishing social network, limited opportunities with social groups, and lack of access to culturally and linguistically relevant health information have all contributed to increased depression among older Asians. In addition, increases in hate speech and racist crimes against Asians have created a hostile living environment for older Asians, further contributing to depression.

Mindfulness-based cognitive therapy (MBCT) is effective for preventing depression relapse and active depression. Our team has created a brief telephone-based MBCT which has been shown to be acceptable primarily white primarily white population. The acceptability of MBCT among older Korean Americans remain understudied.

Community-based organizations (CBOs) are places for accessing federal and state programs, receiving culturally and linguistically appropriate health education, and supporting and socializing with other older Asians. Our preliminary study shows that 1) CBOs are ideal settings for offering MBCT-T because they have the infrastructure, capacity, cultural understanding, and trust of communities, and 2) many CBOs feel the urgency to address older Asians' escalating rates of depression and asked for assistance with training and implementation of MBCT-T.

We will partner with a CBO that serves large older Korean American population to conduct a pilot study to assess the acceptability, feasibility, and preliminary impact of a CBO delivered MBCT program on depression among older Korean Americans.

ELIGIBILITY:
Inclusion Criteria:

* Participants must: (1) self-identify as a Korean person, (2) be between the ages 55 and 89, (3) has mild to moderate depressive symptoms (scores between 5-14 when assessed using Patient Health Questionnaire-9 (PHQ-9), (4) has limited English proficiency (responds "less than very well" when asked "how well do you speak English"?) and fluency in Korean (e.g. able to speak at a native level), and (5) willing to give a written consent to participate in the study.

Exclusion Criteria:

* Individuals will not be able to participate if they have any of the following criteria: (1) major psychiatric diseases that would interfere with participants' ability to participate in or receive the benefit from the mental health interventions (e.g., bipolar disorder, schizophrenia, recent history of psychosis or mania, severe depressive symptoms); (2) used drugs other than those required for medical reasons; (3) serious medical conditions (e.g., poorly controlled diabetes, severe congestive heart failure) that has not been stable for at least 3 months; (4) current active suicidal or self-injurious behavior, potentially necessitating immediate treatment; (5) general conditions that would impede participation in a group intervention (e.g., cognitive impairment, tendencies toward physical aggression); (65) prior history of engaging in formal mindfulness-based interventions including mindfulness-based stress reduction, MBCT, Acceptance and Commitment Therapy, and Dialectical Behavioral Therapy; and (76) significant current meditation practice, specifically more than three hours of insight/mindfulness/Vipassana meditation per week.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ko, MPH,PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not meeting inclusion criteria and other reasons
Period: Overall Study
Arm/Group | Group-based MBCT
Started | 24
Completed Intervention | 22
Completed | 22
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Group-based MBCT
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.58 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: Quick Inventory of Depressive Symptomatology (QIDS-SR); score ranges from 0-27 with higher scores indicating more depressive symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Group-based MBCT
Number analyzed (Participants) | 22
score | 10.29 (4.21)

2. Secondary Outcome: Sleep
Description: Sleep Quality PROMIS measure
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Description: Not different
Arm/Group | Group-based MBCT
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT05965349/Prot_SAP_000.pdf